CLINICAL TRIAL: NCT07048834
Title: Comparison of the Effectiveness of Articaine Local Infusion and Lidocaine Nerve Block in Lower Posterior Tooth Extraction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amjed Fouad Hussein (Other)
Responsible Party: Sponsor-Investigator, Amjed Fouad Hussein, Assistant Lecturer, Ahl al-Bayt University
Organization: Ahl al-Bayt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1419
Record Dates: First submitted 2025-05-21; First posted 2025-07-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients anesthetized by 2 % lidocaine with 1:80,000 adrenaline by inferior alveolar nerve block. (Other): This group of (30 patients) will be anesthetized using 2 % lidocaine with 1:80,000 adrenaline by inferior alveolar nerve block technique, Then patients will wait for five minutes after receiving a local anesthetic injection before extraction could begin.
  After that every tooth's buccal, lingual, mesial, and distal surfaces will be examined using a disposable dental explorer. Then by visual analog scale (VAS) which provides accessible, sensitive, valid, and reliable means to measure a variety of subjective parameters the pain score will be registered during tooth extraction
  Interventions: Other: lidocaine local anesthetic drug
- anesthetized by 4 % articaine with 1:100,000 adrenaline via buccal and lingual infiltration. (Other): This group (of 30 patients) will be anesthetized using 4 % articaine with 1:100,000 adrenaline via buccal and lingual infiltration technique in posterior teeth area. Then patients will wait for five minutes after receiving a local anesthetic injection before extraction could begin.
  After that every tooth's buccal, lingual, mesial, and distal surfaces will be examined using a disposable dental explorer. Then by visual analog scale (VAS) which provides accessible, sensitive, valid, and reliable means to measure a variety of subjective parameters the pain score will be registered during tooth extraction.
  Interventions: Other: articaine local anesthetic drug

INTERVENTIONS:
Other: lidocaine local anesthetic drug — Lidocaine Nerve Block technique
  Arms: patients anesthetized by 2 % lidocaine with 1:80,000 adrenaline by inferior alveolar nerve block.
Other: articaine local anesthetic drug — Articaine Local Infusion technique
  Arms: anesthetized by 4 % articaine with 1:100,000 adrenaline via buccal and lingual infiltration.

SUMMARY:
In this study 60 adult patients will participate and divided into two groups (30 for each). The first group will be anesthetized using 2 % lidocaine with 1:80,000 adrenaline by inferior alveolar nerve block technique, while the second group will be anesthetized using 4 % articaine with 1:100,000 adrenaline via buccal and lingual infiltration technique in posterior teeth area. Then patients will wait for five minutes after receiving a local anesthetic injection before extraction could begin.

After that every tooth's buccal, lingual, mesial, and distal surfaces will be examined using a disposable dental explorer. Then by visual analog scale (VAS) which provides accessible, sensitive, valid, and reliable means to measure a variety of subjective parameters the pain score will be registered during tooth extraction.

Female patients who are breastfeeding or pregnant, those allergic to local anesthetics, lacking full mental ability, currently taking opioids, having an infection at the extraction site, or those under the influence of medicines that alter their perception of pain will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* clinically healthy patients

Exclusion Criteria:

* Breastfeeding or pregnant
* Allergic to local anaesthetics drugs
* Lack full mental ability
* Infection at the extraction site
* Patient who currently taking opioids or under the influence of medicines that alter their perception of pain are not candidates for tooth extraction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | five minutes
  It usually is a horizontal line, 100 mm in length, anchored by word descriptors at each end, for example, that represent the severity of symptoms from 0 "no symptoms" to 10 "very severe symptoms." The patient marks on the line the point that the patient believes represents his or her perception of his or her current state.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahl Al Bayt University, Karbala, Iraq

IPD SHARING:
Plan to Share IPD: No
Due to lack of participant consent for data Sharing. so, Individual participant data will not be shared due to the absence of specific provisions for broad external data sharing within the original informed consent documents signed by participants. Retrospective consent for such sharing is not feasible for this study population.

REFERENCES:
- [Background] Webster S Jr, Drum M, Reader A, Fowler S, Nusstein J, Beck M. How Effective Is Supplemental Intraseptal Anesthesia in Patients with Symptomatic Irreversible Pulpitis? J Endod. 2016 Oct;42(10):1453-7. doi: 10.1016/j.joen.2016.07.002. PMID 27663614
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22822998/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34395896/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28127498/